CLINICAL TRIAL: NCT07129395
Title: Optimizing Measurement of Anticoagulation Adherence
Brief Title: Anticoagulation Adherence Measurement Strategies
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: Anticoagulation Adherence; H30MC24047 (Other Grant/Funding Number: Health Resources and Service Administration)
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Anticoagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Single center study to evaluate the feasibility of using 3 different strategies to measure adherence among children, adolescents, and young adults prescribed an anticoagulation medication

DETAILED DESCRIPTION:
This is an observational study with a maximum of 5 study visits during the 12-week study period. The study visit schedule has been designed to align with current clinical care practices. Adherence will be assessed via the EAMDs device, as well as by self-report measure in the BAT and by staff telephone inquiry regarding pharmacy refill data. Adherence data will be used to compute rates and trajectories of adherence to anticoagulants.

It is anticipated that this study will conclude in approximately 2 years, including data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Anticoagulated CCHMC patients ages 0 to 29.9 years and their caregivers (where applicable for patients < 18 years)
* Able to provide informed consent
* Duration of anticoagulation planned for the outpatient setting is 4 weeks or longer
* Willing and able to participate in telephone and in person study visits
* For patients < 18 years, both patient and caregiver agree to participate

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Duration of anticoagulation is planned for < 4 weeks in the outpatient setting
* Anticoagulant drug will not fit into the EAMD
* Unable to participate in telephone study visit

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric, adolescents and young adults prescribed an anticoagulation medication.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2026-10-04 (Estimated)

PRIMARY OUTCOMES:
Measure adherence via electronic adherence monitoring device (EAMD) | 12 weeks
  Participants will be provided with a MEMS® Cap if they are prescribed an oral medication and a MEMS® Injectable if they are prescribed an injectable medication. Patients and families will then be trained by study nurse coordinator (NC) or principal investigator (PI) regarding how to use the MEMS® for medication administration throughout the study.

SECONDARY OUTCOMES:
Rate barriers to adherence. | 12 weeks
  Characterize the rate of barriers to adherence in a sample of children and adolescents and young adults prescribed anticoagulants using data from three different adherence measurements.
Self-reported barriers to adherence. | 12 weeks
  Characterize the self-reported barriers to adherence in a sample of children and adolescents and young adults prescribed anticoagulants using data from three different adherence measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Luchtman-Jones, MD, Principal Investigator — Region V-East Great Lake Region, Cincinnati Children's Hospital Medical Center, University of Cincinnati College of Medicine
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Andrew M, David M, Adams M, Ali K, Anderson R, Barnard D, Bernstein M, Brisson L, Cairney B, DeSai D, et al. Venous thromboembolic complications (VTE) in children: first analyses of the Canadian Registry of VTE. Blood. 1994 Mar 1;83(5):1251-7. PMID 8118029
- [Background] Gibson BES, Chalmers EA et al. Thromboembolism in childhood: a prospective 2-year BPSU study in the United Kingdom. February 2001-February 2003. Br J Haematol. 2004;1:OC422
- [Background] van Ommen CH, Heijboer H, Buller HR, Hirasing RA, Heijmans HS, Peters M. Venous thromboembolism in childhood: a prospective two-year registry in The Netherlands. J Pediatr. 2001 Nov;139(5):676-81. doi: 10.1067/mpd.2001.118192. PMID 11713446
- [Background] Raffini L, Huang YS, Witmer C, Feudtner C. Dramatic increase in venous thromboembolism in children's hospitals in the United States from 2001 to 2007. Pediatrics. 2009 Oct;124(4):1001-8. doi: 10.1542/peds.2009-0768. Epub 2009 Sep 7. PMID 19736261
- [Background] Kerlin BA. Current and future management of pediatric venous thromboembolism. Am J Hematol. 2012 May;87 Suppl 1(0 1):S68-74. doi: 10.1002/ajh.23131. Epub 2012 Feb 24. PMID 22367975
- [Background] Monagle P, Newall F. Management of thrombosis in children and neonates: practical use of anticoagulants in children. Hematology Am Soc Hematol Educ Program. 2018 Nov 30;2018(1):399-404. doi: 10.1182/asheducation-2018.1.399. PMID 30504338
- [Background] Monagle P, Chan AKC, Goldenberg NA, Ichord RN, Journeycake JM, Nowak-Gottl U, Vesely SK. Antithrombotic therapy in neonates and children: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e737S-e801S. doi: 10.1378/chest.11-2308. PMID 22315277
- [Background] Luchtman-Jones L. Venous thromboembolism and anticoagulation safety: who is watching the children? Pediatr Blood Cancer. 2014 Nov;61(11):1916-7. doi: 10.1002/pbc.25145. Epub 2014 Jul 22. No abstract available. PMID 25053292
- [Background] Jones S, McLoughlin S, Piovesan D, Savoia H, Monagle P, Newall F. Safety and Efficacy Outcomes of Home and Hospital Warfarin Management Within a Pediatric Anticoagulation Clinic. J Pediatr Hematol Oncol. 2016 Apr;38(3):216-20. doi: 10.1097/MPH.0000000000000502. PMID 26808370
- [Background] Simons LE, Blount RL. Identifying barriers to medication adherence in adolescent transplant recipients. J Pediatr Psychol. 2007 Aug;32(7):831-44. doi: 10.1093/jpepsy/jsm030. Epub 2007 May 23. PMID 17522111
- [Background] Modi AC, Pai AL, Hommel KA, Hood KK, Cortina S, Hilliard ME, Guilfoyle SM, Gray WN, Drotar D. Pediatric self-management: a framework for research, practice, and policy. Pediatrics. 2012 Feb;129(2):e473-85. doi: 10.1542/peds.2011-1635. Epub 2012 Jan 4. PMID 22218838
- [Background] Rapoff M. Adherence to pediatric medical regimens. 2nd ed. Issues in Clinical Child Psychology. New York, NY: Springer Science+Business Media; 2010
- [Background] Bhatia S, Landier W, Hageman L, Kim H, Chen Y, Crews KR, Evans WE, Bostrom B, Casillas J, Dickens DS, Maloney KW, Neglia JP, Ravindranath Y, Ritchey AK, Wong FL, Relling MV. 6MP adherence in a multiracial cohort of children with acute lymphoblastic leukemia: a Children's Oncology Group study. Blood. 2014 Oct 9;124(15):2345-53. doi: 10.1182/blood-2014-01-552166. Epub 2014 May 14. PMID 24829202
- [Background] Wu YP, Stenehjem DD, Linder LA, Yu B, Parsons BG, Mooney R, Fluchel MN. Adherence to Oral Medications During Maintenance Therapy Among Children and Adolescents With Acute Lymphoblastic Leukemia: A Medication Refill Analysis. J Pediatr Oncol Nurs. 2018 Mar/Apr;35(2):86-93. doi: 10.1177/1043454217741877. Epub 2017 Nov 30. PMID 29188741
- [Background] Quittner AL, Modi AC, Lemanek KL, Ievers-Landis CE, Rapoff MA. Evidence-based assessment of adherence to medical treatments in pediatric psychology. J Pediatr Psychol. 2008 Oct;33(9):916-36; discussion 937-8. doi: 10.1093/jpepsy/jsm064. Epub 2007 Sep 10. PMID 17846042
- [Background] Vrijens B, Antoniou S, Burnier M, de la Sierra A, Volpe M. Current Situation of Medication Adherence in Hypertension. Front Pharmacol. 2017 Mar 1;8:100. doi: 10.3389/fphar.2017.00100. eCollection 2017. PMID 28298894
- [Background] Riekert KA, Rand CS. Electronic monitoring of medication adherence: When is high-tech best? J Clin Psychol Med Settings. 2002;9:25-34
- [Background] Chan AH, Harrison J, Black PN, Mitchell EA, Foster JM. Using electronic monitoring devices to measure inhaler adherence: a practical guide for clinicians. J Allergy Clin Immunol Pract. 2015 May-Jun;3(3):335-49.e1-5. doi: 10.1016/j.jaip.2015.01.024. Epub 2015 Apr 1. PMID 25840665
- [Background] McGrady ME, Holbein CE, Smith AW, Morrison CF, Hommel KA, Modi AC, Pai ALH, Ramsey RR. An Independent Evaluation of the Accuracy and Usability of Electronic Adherence Monitoring Devices. Ann Intern Med. 2018 Sep 18;169(6):419-422. doi: 10.7326/M17-3306. Epub 2018 May 22. No abstract available. PMID 29800004
- [Background] McGrady ME, Ramsey RR. Using Electronic Monitoring Devices to Assess Medication Adherence: a Research Methods Framework. J Gen Intern Med. 2020 Sep;35(9):2707-2714. doi: 10.1007/s11606-020-05905-z. Epub 2020 May 21. PMID 32440997
- [Background] Nieuwlaat R, Wilczynski N, Navarro T, Hobson N, Jeffery R, Keepanasseril A, Agoritsas T, Mistry N, Iorio A, Jack S, Sivaramalingam B, Iserman E, Mustafa RA, Jedraszewski D, Cotoi C, Haynes RB. Interventions for enhancing medication adherence. Cochrane Database Syst Rev. 2014 Nov 20;2014(11):CD000011. doi: 10.1002/14651858.CD000011.pub4. PMID 25412402
- [Background] De Bleser L, De Geest S, Vandenbroeck S, Vanhaecke J, Dobbels F. How accurate are electronic monitoring devices? A laboratory study testing two devices to measure medication adherence. Sensors (Basel). 2010;10(3):1652-60. doi: 10.3390/s100301652. Epub 2010 Mar 2. PMID 22294891